CLINICAL TRIAL: NCT03785470
Title: Vascular and Metabolic Consequences of Adopting a Westernized Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Camila Manrique, Associate Professor, Endocrinology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012869
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Vascular Diseases
Keywords: arterial stiffness; endothelial dysfunction; fructose; physical inactivity
MeSH Terms: conditions — Vascular Diseases; Sedentary Behavior | interventions — Fructose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fructose and physical inactivity (Experimental): Subjects will consume 6 cans of soda per day and restrict their physical activity.
  Interventions: Other: Fructose and physical inactivity

INTERVENTIONS:
Other: Fructose and physical inactivity — Subjects will drink 6 cans of regular sodas daily (divided throughout the day) and will decreased physical activity to less than 5000 steps daily for 10 days.

SUMMARY:
The purpose of this study is to determine if short-term adoption of a Westernized lifestyle characterized by physical inactivity and increased consumption of fructose will result in metabolic and vascular dysfunction. Healthy individuals aged 18-45 years old will undergo an acute period of physical inactivity (10 days) coupled with increased fructose consumption. Augmented fructose consumption will be achieved via commercially available soda beverages which are high in fructose. Vascular and metabolic function measures will be performed before and after the 10-day intervention.

DETAILED DESCRIPTION:
Men and women who regularly engage in >10,000 steps per day, age 18-45 years, body mass index < 30 kg/m2, and with no history of chronic disease will be recruited. Subjects who are eligible will undergo an acute period of physical inactivity (10 days) coupled with increased fructose consumption (6 cans/day). Physical activity levels will be assessed via a pedometer to quantify if individuals achieve <5000 steps/day. Vascular and metabolic function measures will be performed before and after the 10-day intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who regularly engage in >10,000 steps per day
* Age 18-45 years
* Body mass index < 30 kg/m2
* No history of chronic disease

Exclusion Criteria:

* Known cardiovascular disease including hypertension, heart failure, coronary artery disease, and stroke
* Renal or hepatic diseases
* Active cancer
* Autoimmune diseases
* Current use of immunosuppressant therapy
* Excessive alcohol consumption (> 14 drinks/week for men and >7 drinks/week for women)
* Current tobacco use
* Current pregnancy
* Diagnosis of type 2 diabetes
* Regular consumption of >2 non-diet sodas/day

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Change in Insulin-stimulated leg blood flow | this will be assessed at baseline and at the final visit (10 days)
  Subjects will be instrumented with EKG for contrast-enhanced ultrasound (CEU) measurements. We will perform a hyperinsulinemic euglycemic clamp to evaluate microvascular perfusion of skeletal muscle via CEU. Insulin will be infused at a constant rate to mimic postprandial insulin concentrations and glucose maintained at fasting values via a variable 20% dextrose infusion. At baseline and in the steady state phase of the insulin clamp, we will assess microvascular perfusion in the vastus lateralis muscle using CEU (IE-33, Philips Ultrasound), via infusion of perflutren lipid microspheres. Microvascular perfusion will be assessed as an A-value. A is the video intensity plateau after complete replenishment reflecting relative microvascular blood volume (MBV).

SECONDARY OUTCOMES:
Change in Brachial artery flow mediated dilation (FMD) | this will be assessed at baseline and at the final visit (10 days)
  Brachial artery FMD will be assessed at baseline and at 10 days. FMD is a measurement of conduit artery endothelial function. FMD is assessed immediately after each PWV measurement. Shear rate AUC until peak diameter is calculated as stimulus for FMD and used in covariate analysis. All measurements will be performed by the same technician.
Change in carotid femoral pulse wave velocity (cfPWV) | this will be assessed at baseline and at the final visit (10 days)
  It is the gold standard non-invasive index of arterial stiffness. Transit time between carotid and femoral pressure waves is calculated using the foot-to-foot method. cfPWV is calculated as distance traveled by the pulse wave (i.e., femoral location-sternal notch minus sternal notch-carotid location) divided by pulse transit time. All the measurements will be done by the same technician

CONTACTS AND LOCATIONS:
Overall Officials: Camila Manrique Acevedo, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No